CLINICAL TRIAL: NCT00005021
Title: Phase I Evaluation of Topotecan in Combination With Paclitaxel and Carboplatin
Brief Title: Combination Chemotherapy With or Without Biological Therapy in Treating Patients With Refractory Solid Tumor or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FCCC-96004; CDR0000064913 (Registry Identifier: PDQ (Physician Data Query)); NCI-T95-0075H (Other Grant/Funding Number: National Cancer Institute)
Record Dates: First submitted 2000-04-06; First posted 2004-05-03 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Lymphoma; Small Intestine Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; recurrent adult Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; small intestine lymphoma; unspecified adult solid tumor, protocol specific; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; recurrent adult T-cell leukemia/lymphoma; primary central nervous system non-Hodgkin lymphoma; AIDS-related peripheral/systemic lymphoma; AIDS-related primary CNS lymphoma; intraocular lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; angioimmunoblastic T-cell lymphoma; anaplastic large cell lymphoma; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; recurrent mycosis fungoides/Sezary syndrome; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Intraocular Lymphoma; Lymphoma, Mantle-Cell; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Mycosis Fungoides; Sezary Syndrome; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Filgrastim; Carboplatin; Paclitaxel; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: filgrastim
Drug: carboplatin
Drug: paclitaxel
Drug: topotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug, giving the drugs in different ways, and combining biological therapy with chemotherapy may kill more cancer cells.

PURPOSE: Phase I trial to study the effectiveness of topotecan, paclitaxel, and carboplatin with or without filgrastim in treating patients who have advanced solid tumor or lymphoma that has not responded to standard therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated doses of combined topotecan, paclitaxel, and carboplatin (TOPO/TAX/CBDCA) with or without filgrastim (G-CSF) in patients with advanced solid tumors or lymphomas. II. Determine the toxic effects of this regimen in these patients. III. Determine the pharmacokinetics of TOPO/TAX/CBDCA and whether TAX/CBDCA will affect the pharmacokinetics of TOPO on day 1 as compared to TOPO administered alone on day 3. IV. Describe any clinical responses observed in these patients.

OUTLINE: This is a dose escalation study of the combination topotecan/paclitaxel/carboplatin. Patients are stratified according to prior chemotherapy and radiotherapy (yes vs no). Part I: Patients receive topotecan IV on days 1-3 and paclitaxel IV over 3 hours and carboplatin IV over 30-60 minutes, on day 1. Part II: Patients receive topotecan, paclitaxel, and carboplatin as in part I, plus filgrastim (G-CSF) on days 6-19. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity Cohorts of 3-6 patients receive escalating doses of topotecan/paclitaxel/carboplatin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicity.

PROJECTED ACCRUAL: Approximately 20-30 patients will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven advanced solid tumor or lymphoma that is refractory to standard therapy or for which no standard therapy exists or for which the drugs used in this regimen constitute standard therapy Brain metastasis eligible provided: Evidence of neurologic improvement or normalization No evidence of radiographic progression after appropriate therapy Steroid dose stable (if given)

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0 or 1 Life expectancy: Greater than 3 months Hematopoietic: Absolute granulocyte count at least 2,000/mm2 Platelet count at least 100,000/mm2 Hepatic: Bilirubin no greater than 1.5 mg/dL Transaminases less than 3 times normal Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance at least 60 mL/min Cardiovascular: No myocardial infarction within 6 months No history of congestive heart failure No uncontrolled angina No uncontrolled arrhythmia Other: No concurrent medical illness or active infection that would render treatment unsafe Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Prior topotecan, paclitaxel, and carboplatin allowed if progression observed greater than 3 months after last dose No prior mitomycin or nitrosoureas No more than 1 prior chemotherapy regimen At least 4 weeks since chemotherapy and recovered (alopecia allowed) Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy to more than 25% of bone marrow At least 4 weeks since radiotherapy and recovered (alopecia allowed) Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 1996-07; Primary Completion 2003-05 (Actual); Study Completion 2003-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corey J. Langer, MD, Study Chair — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States